CLINICAL TRIAL: NCT05127538
Title: Assessment of Balance and Gait in Patients With Diabetic Peripheral Neuropathy
Brief Title: Balance and Gait in Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozlem Yuruk, Assoc. Prof., Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KA21/317
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Neuropathy, Diabetic; Pain, Neuropathic; Gait Disorder, Sensorimotor
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia; Gait Disorders, Neurologic | interventions — Gait Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individuals diagnosed with neuropathic pain due to type 2 diabetes (Active Comparator): * Individuals between the ages of 40-65
  * Individuals who take 4 points or more from the Douleur Neuropathique en 4 questions (DN4) questionnaire
  * Individuals who take 12 points or more from the Leeds Assessment of Neuropathic Signs and Symptoms (LANSS) scale
  Interventions: Diagnostic Test: Gait analysis; Diagnostic Test: Balance Assessment
- Individuals with type 2 diabetes but no neuropathic pain (Active Comparator): * Individuals between the ages of 40-65
  * Individuals who take 4 points from the Douleur Neuropathique en 4 questions (DN4) questionnaire
  * Individuals who take 12 points from the Leeds Assessment of Neuropathic Signs and Symptoms (LANSS) scale
  Interventions: Diagnostic Test: Gait analysis; Diagnostic Test: Balance Assessment
- Healthy control group (Active Comparator): * Individuals between the ages of 40-65
  * Individuals who have no pain (Taking 1 point or less according to the Visual Pain Scale)
  Interventions: Diagnostic Test: Gait analysis; Diagnostic Test: Balance Assessment

INTERVENTIONS:
Diagnostic Test: Gait analysis — Gait analysis Zebris Rehawalk (Zebris Medical GmbH, Germany) computerized gait evaluation system is used to assess the kinetic and kinematic analysis of the gait. The system consists of a treadmill and a computer. For gait assessment, patients walk at their preferred comfortable walking speed.
Diagnostic Test: Balance Assessment — Static and dynamic balance Static and dynamic balance and stability limit values are evaluated with the E-LINK FP3 Force Plate (Biometrics Ltd, United Kingdom) system. The device consists of a computer and a platform on which individuals can place their feet. For static balance measurement, individuals are asked to place their feet on the marked places on the platform and hold an object on the computer screen at a fixed point for 30 seconds without support from their hands. For dynamic balance, individuals need to follow a moving object on the computer screen for 30 seconds by putting their body weight forward, backward, and sideways with their feet.

SUMMARY:
The aim of the study is to evaluate the effects of neuropathic pain due to type 2 diabetes on balance and gait. The study is a prospective controlled study. The study is being carried out at the Physical Therapy and Rehabilitation Center Gait Analysis Laboratory Unit in Turkey.

Individuals diagnosed with neuropathic pain due to Type 2 Diabetes and individuals with diabetes without neuropathic pain are included in the study by clinical examination and tests by a physician. At the same time, healthy individuals are participating as the control group.

There will 3 groups in the study :

Group 1: Individuals diagnosed with neuropathic pain due to type 2 diabetes (n=14) Group 2: Individuals with type 2 diabetes but no neuropathic pain (n=14) Group 3: Healthy control group (n=14)

Assessments:

Individual and clinical characteristics of individuals: age, gender, height, body weight, marital status, education level, duration of complaints, and dominant side.

Douleur Neuropathique en 4 questions (DN4) Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Pain Questionnaire Visual Analog Scale (VAS) Gait analysis Static and dynamic balance

The data will be analyzed using the statistical program for social sciences (SPSS) version 21.0 (IBM SPSS Statistics for Windows, Armonk, NY: IBM Corp.). The data will be expressed as mean standard deviation (X±SD) and number (n%). The homogeneity of the groups will be evaluated with the Levene Test. Balance, plantar pressure, and walking values between the groups will be compared using the Kruskal Wallis Test. All the statistical analyses will be set a priori at an alpha level of p<0.05.

DETAILED DESCRIPTION:
Diabetes is a metabolic disorder characterized by chronic hyperglycemia due to a deficiency in the insulin hormone. The most common symptoms of type 2 diabetes include diabetic peripheral neuropathy, which results in hyperglycemia, polyuria, muscle weakness, numbness, and tingling sensations in the extremities.

Diabetic peripheral neuropathy, one of the most common long-term complications of diabetes, is characterized by damage to sensory and motor nerve fibers caused by uncontrolled hyperglycemia, seen in approximately 50% of diabetic patients. In diabetic peripheral neuropathy, there is an impairment in the conduction of afferent and efferent fibers. Thus, decreased muscle strength, weakening in postural control, and tactile sensation loss occurs compared to healthy individuals.

Pain is one of the most common problems in diabetic peripheral neuropathy. Pain and paresthesia increase especially at night in the lower extremities. Diabetic neuropathic pain results in different physical problems such as the increased risk of falling, loss of balance and coordination while standing or walking, susceptibility to injuries due to sensory loss, sleep disorders, and fatigue.

Gait disorders are one of the complications seen in diabetic peripheral neuropathy. Neuromuscular damage due to neuropathy causes alterations in the biomechanics of the lower extremities, and thus, deterioration in the time-distance characteristics of gait such as stride length, stride width, double and single support period.

Studies report that increased dynamic mediolateral and anteroposterior swing cause postural instability. Falls caused by lack of postural control and gait disorders are 15 times more common in patients with diabetic peripheral neuropathy than in healthy individuals. Therefore, it is necessary to evaluate the balance and calculate the risk of falling.

In the literature, although studies are examining kinetic analyzes of gait in patients with diabetic neuropathy, few studies were evaluating kinematic analyzes and stability limits. In addition, the balance and gait parameters of patients with neuropathy were compared with healthy individuals in studies, but no study compared with diabetic patients without neuropathy. Therefore, the aim of the study is to evaluate the effects of neuropathic pain due to type 2 diabetes on balance and gait.

METHODS The study is a prospective controlled study. The study is being carried out at the Physical Therapy and Rehabilitation Center Gait Analysis Laboratory Unit in Ankara-Turkey. Individuals diagnosed with neuropathic pain due to Type 2 Diabetes and individuals with diabetes without neuropathic pain are included in the study by clinical examination and tests by a physician. At the same time, healthy individuals are participating as the control group.

The groups will:

Group 1: Individuals diagnosed with neuropathic pain due to type 2 diabetes (n=14) Group 2: Individuals with type 2 diabetes but no neuropathic pain (n=14) Group 3: Healthy control group (n=14) A written informed consent form is being obtained from all individuals.

Inclusion criteria for individuals with neuropathic pain due to type 2 diabetes:

* Being between the ages of 40-65
* Taking 4 points or more from the Douleur Neuropathique en 4 questions (DN4) questionnaire
* Taking 12 points or more from the Leeds Assessment of Neuropathic Signs and Symptoms (LANSS) scale

Inclusion criteria for individuals with type 2 diabetes but no neuropathic pain:

* Being between the ages of 40-65
* Taking below 4 points from the Douleur Neuropathique en 4 questions (DN4) questionnaire
* Taking below 12 points from the Leeds Assessment of Neuropathic Signs and Symptoms (LANSS) scale

Inclusion criteria of healthy individuals in the study:

* Being between the ages of 40-65
* Have no pain (Taking 1 point or less according to the Visual Pain Scale)

Exclusion criteria:

* Having a complaint of pain from different etiology
* Having a diabetic foot ulcer
* Presence of neurological disease that may cause central neuropathic pain such as stroke, traumatic brain injury, multiple sclerosis
* Had orthopedic surgery in the last six months
* Having vision problems related to diabetes
* Had a diagnosis of vestibular disorders (Bening Paroxysmal Positional Vertigo, Meniere's Disease, etc.)
* Having chronic pain syndrome such as Fibromyalgia Syndrome

Assessments

Information Form:

The researchers record individual and clinical characteristics of individuals such as age, gender, height, body weight, marital status, education level, duration of complaints, and dominant side.

Douleur Neuropathique en 4 questions (DN4):

DN4 is a scale consisting of 10 questions evaluating neuropathic pain. Seven items are related to pain symptoms and three items include a clinical examination. The scale asks whether patients have burning, painful cold, electric shock, tingling, prickling, numbness, and itching. In addition, sensory changes in the patient are examined with cotton, pins, and brushing. While 1 point is given for each item in scoring, a score of 4 or more indicates the presence of neuropathic pain. Taking 4 points or more from the DN4 is one of the criteria for identifying neuropathic pain in the study.

Leeds Assessment of Neuropathic Symptoms and Signs (LANSS):

The LANSS is a validated questionnaire that consists of 7 items, can distinguish neuropathic pain from nociceptive pain, and is easy to score in clinical settings. The first part of the scale consists of 5 items questioning the pain symptoms and answered as yes or no. The patient is asked to think about the pain he or she has felt during the past week. In the second part, the presence of allodynia and the sharp-blunt threshold value is evaluated by sensory examination. The questionnaire is calculated between 0-24 points. Twelve points and above indicates neuropathic pain. Taking below 12 points from the LANSS scale is one of the criteria for identifying neuropathic pain in the study.

Visual Analog Scale (VAS):

VAS is a scale that evaluates pain on a horizontal 100 mm line. On the line, the left side indicates 'no pain' and the right side indicates 'the most severe pain imaginable. Healthy individuals are asked to mark a point on the line according to the severity of the pain they feel.

Gait analysis:

Zebris Rehawalk (Zebris Medical GmbH, Germany) computerized gait evaluation system is used to assess the kinetic and kinematic analysis of the gait. The dynamic foot pressure distribution is also analyzed with the pedobarography integrated into this system. The system consists of a treadmill and a computer. For gait assessment, patients walk at their preferred comfortable walking speed. In the evaluation, joint angles, walking speed, step lengths,right-left and anterior-posterior weight transfer, left-right foot rotation, lateral mobility, the center of gravity movement, and swing area are recorded. Evaluation time is approximately 5 minutes.

Balance:

Static and dynamic balance and stability limit values are evaluated with the E-LINK FP3 Force Plate (Biometrics Ltd, United Kingdom) system. For static balance measurement, individuals are asked to place their feet on the marked places on the platform and hold an object on the computer screen at a fixed point for 30 seconds without support from their hands. For dynamic balance, individuals need to follow a moving object on the computer screen for 30 seconds by putting their body weight forward, backward, and sideways with their feet. The device gives the balance value as a printout by calculating the deviation rate of the individual from the target and the risk of falling forward, backward, and sideways. The measurement takes an average of 10 minutes.

Statistical Analysis For the sample size calculation G*Power Ver. 3.0.10 (Franz Faul, Universität Kiel, Germany) was used. Step length is the primer outcome of the study from the reference article. The analysis was carried out with an effective width of f=0.59, a power of 90%, and a margin of error of 0.05. It was found that 14 individuals in all three groups and a total of 42 individuals should be included in the study.

The data of the study will be analyzed by using the Statistical Program for Social Sciences (SPSS) version 23.0 (IBM SPSS Statistics for Windows, Armonk, NY: IBM Corp.). Descriptive data will be given as mean and standard deviation if numerical variables provide the parametric assumption, if not, median and minimum-maximum values will be given. Qualitative variables will be given with frequency and percentage values. Kruskal Wallis Test will be used for the comparison of independent samples. All the statistical analyses will be set a priori at an alpha level of p<0.05

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for individuals with neuropathic pain due to type 2 diabetes:

* Being between the ages of 40-65
* Taking 4 points or more from the Douleur Neuropathique en 4 questions (DN4) questionnaire
* Taking 12 points or more from the Leeds Assessment of Neuropathic Signs and Symptoms (LANSS) scale

Inclusion criteria for individuals with type 2 diabetes but no neuropathic pain:

* Being between the ages of 40-65
* Taking below 4 points from the Douleur Neuropathique en 4 questions (DN4) questionnaire
* Taking below 12 points from the Leeds Assessment of Neuropathic Signs and Symptoms (LANSS) scale

Inclusion criteria of healthy individuals in the study:

* Being between the ages of 40-65
* Have no pain (Taking 1 point or less according to the Visual Pain Scale)

Exclusion Criteria:

* Having a complaint of pain from different etiology
* Having a diabetic foot ulcer
* Presence of neurological disease that may cause central neuropathic pain such as stroke, traumatic brain injury, multiple sclerosis
* Had orthopedic surgery in the last six months
* Having vision problems related to diabetes
* Had a diagnosis of vestibular disorders (Bening Paroxysmal Positional Vertigo, Meniere's Disease, etc.)
* Having chronic pain syndrome such as Fibromyalgia Syndrome

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Step Length | 5 minutes
  Zebris Rehawalk (Zebris Medical GmbH, Germany) computerized gait evaluation system is used to assess the kinetic and kinematic analysis of the gait. The dynamic foot pressure distribution is analyzed with the pedobarography integrated into this system. The system consists of a treadmill and a computer. While the computer automatically detects the patient's hip, knee, and ankle, measures an individual's foot pressure on the ground. For gait assessment, patients walk at their preferred comfortable walking speed.
Gait velocity | 5 minutes
  Zebris Rehawalk (Zebris Medical GmbH, Germany) computerized gait evaluation system is used to assess the kinetic and kinematic analysis of the gait. The dynamic foot pressure distribution is analyzed with the pedobarography integrated into this system. The system consists of a treadmill and a computer. While the computer automatically detects the patient's hip, knee, and ankle, measures an individual's foot pressure on the ground. For gait assessment, patients walk at their preferred comfortable walking speed.
cadance | 5 minutes
  Zebris Rehawalk (Zebris Medical GmbH, Germany) computerized gait evaluation system is used to assess the kinetic and kinematic analysis of the gait. The dynamic foot pressure distribution is analyzed with the pedobarography integrated into this system. The system consists of a treadmill and a computer. While the computer automatically detects the patient's hip, knee, and ankle, measures an individual's foot pressure on the ground. For gait assessment, patients walk at their preferred comfortable walking speed.
Foot pressure distribution | 5 minutes
  Zebris Rehawalk (Zebris Medical GmbH, Germany) computerized gait evaluation system is used to assess the kinetic and kinematic analysis of the gait. The dynamic foot pressure distribution is analyzed with the pedobarography integrated into this system. The system consists of a treadmill and a computer. While the computer automatically detects the patient's hip, knee, and ankle, measures an individual's foot pressure on the ground. For gait assessment, patients walk at their preferred comfortable walking speed.
static balance | 5 minutes
  Static and dynamic balance and stability limit values are evaluated with the E-LINK FP3 Force Plate (Biometrics Ltd, United Kingdom) system. The device consists of a computer and a platform on which individuals can place their feet. For static balance measurement, individuals are asked to place their feet on the marked places on the platform and hold an object on the computer screen at a fixed point for 30 seconds without support from their hands. The device gives the balance value as a printout by calculating the deviation rate of the individual from the target and the risk of falling forward, backward, and sideways.
Dynamic Balance | 5 minutes
  Static and dynamic balance and stability limit values are evaluated with the E-LINK FP3 Force Plate (Biometrics Ltd, United Kingdom) system. The device consists of a computer and a platform on which individuals can place their feet. For dynamic balance, individuals need to follow a moving object on the computer screen for 30 seconds by putting their body weight forward, backward, and sideways with their feet. The device gives the balance value as a printout by calculating the deviation rate of the individual from the target and the risk of falling forward, backward, and sideways.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Yuruk, Assoc.Prof, Study Director — Baskent University; Suleyman Korkusuz, MSc, Principal Investigator — Hacettepe University
Locations (3):
- Turkey (Türkiye) (3):
  - Hacettepe University, Ankara
  - Baskent University, Ankara
  - Fizyocare Rehabilitation Center, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anjos DM, Gomes LP, Sampaio LM, Correa JC, Oliveira CS. Assessment of plantar pressure and balance in patients with diabetes. Arch Med Sci. 2010 Mar 1;6(1):43-8. doi: 10.5114/aoms.2010.13506. Epub 2010 Mar 9. PMID 22371719
- [Background] Awotidebe TO, Ativie RN, Oke KI, Akindele MO, Adedoyin RA, Olaogun MO, Olubayode TE, Kolawole BA. Relationships among exercise capacity, dynamic balance and gait characteristics of Nigerian patients with type-2 diabetes: an indication for fall prevention. J Exerc Rehabil. 2016 Dec 31;12(6):581-588. doi: 10.12965/jer.1632706.353. eCollection 2016 Dec. PMID 28119881
- [Background] Huang CK, Shivaswamy V, Thaisetthawatkul P, Mack L, Stergiou N, Siu KC. An altered spatiotemporal gait adjustment during a virtual obstacle crossing task in patients with diabetic peripheral neuropathy. J Diabetes Complications. 2019 Feb;33(2):182-188. doi: 10.1016/j.jdiacomp.2018.10.005. Epub 2018 Oct 17. PMID 30442545
- [Background] Simmons RW, Richardson C, Pozos R. Postural stability of diabetic patients with and without cutaneous sensory deficit in the foot. Diabetes Res Clin Pract. 1997 Jun;36(3):153-60. doi: 10.1016/s0168-8227(97)00044-2. PMID 9237781
- [Background] Tapp RJ, Shaw JE, de Courten MP, Dunstan DW, Welborn TA, Zimmet PZ; AusDiab Study Group. Foot complications in Type 2 diabetes: an Australian population-based study. Diabet Med. 2003 Feb;20(2):105-13. doi: 10.1046/j.1464-5491.2003.00881.x. PMID 12581261
- [Background] Lafond D, Corriveau H, Prince F. Postural control mechanisms during quiet standing in patients with diabetic sensory neuropathy. Diabetes Care. 2004 Jan;27(1):173-8. doi: 10.2337/diacare.27.1.173. PMID 14693985
- [Background] Allet L, Armand S, Aminian K, Pataky Z, Golay A, de Bie RA, de Bruin ED. An exercise intervention to improve diabetic patients' gait in a real-life environment. Gait Posture. 2010 Jun;32(2):185-90. doi: 10.1016/j.gaitpost.2010.04.013. Epub 2010 May 14. PMID 20471273
- [Background] Dyck PJ, Overland CJ, Low PA, Litchy WJ, Davies JL, Dyck PJ, O'Brien PC; Cl vs. NPhys Trial Investigators; Albers JW, Andersen H, Bolton CF, England JD, Klein CJ, Llewelyn JG, Mauermann ML, Russell JW, Singer W, Smith AG, Tesfaye S, Vella A. Signs and symptoms versus nerve conduction studies to diagnose diabetic sensorimotor polyneuropathy: Cl vs. NPhys trial. Muscle Nerve. 2010 Aug;42(2):157-64. doi: 10.1002/mus.21661. PMID 20658599
- [Background] Barrett AM, Lucero MA, Le T, Robinson RL, Dworkin RH, Chappell AS. Epidemiology, public health burden, and treatment of diabetic peripheral neuropathic pain: a review. Pain Med. 2007 Sep;8 Suppl 2:S50-62. doi: 10.1111/j.1526-4637.2006.00179.x. PMID 17714116
- [Background] Higgins DM, Heapy AA, Buta E, LaChappelle KM, Serowik KL, Czlapinski R, Kerns RD. A randomized controlled trial of cognitive behavioral therapy compared with diabetes education for diabetic peripheral neuropathic pain. J Health Psychol. 2022 Mar;27(3):649-662. doi: 10.1177/1359105320962262. Epub 2020 Oct 19. PMID 33070667
- [Background] Izgu N, Gok Metin Z, Karadas C, Ozdemir L, Metinarikan N, Corapcioglu D. Progressive Muscle Relaxation and Mindfulness Meditation on Neuropathic Pain, Fatigue, and Quality of Life in Patients With Type 2 Diabetes: A Randomized Clinical Trial. J Nurs Scholarsh. 2020 Sep;52(5):476-487. doi: 10.1111/jnu.12580. Epub 2020 Jun 13. PMID 32536026
- [Background] Gok Metin Z, Arslan IE. Diabetic Peripheral Neuropathic Pain From the Perspective of Turkish Patients: A Qualitative Study. J Transcult Nurs. 2018 Nov;29(6):514-522. doi: 10.1177/1043659617753044. Epub 2018 Jan 17. PMID 29338623
- [Background] Allet L, Armand S, de Bie RA, Golay A, Pataky Z, Aminian K, de Bruin ED. Clinical factors associated with gait alterations in diabetic patients. Diabet Med. 2009 Oct;26(10):1003-9. doi: 10.1111/j.1464-5491.2009.02811.x. PMID 19900232
- [Background] Almurdhi MM, Brown SJ, Bowling FL, Boulton AJM, Jeziorska M, Malik RA, Reeves ND. Altered walking strategy and increased unsteadiness in participants with impaired glucose tolerance and Type 2 diabetes relates to small-fibre neuropathy but not vitamin D deficiency. Diabet Med. 2017 Jun;34(6):839-845. doi: 10.1111/dme.13316. Epub 2017 Feb 9. PMID 28103405
- [Background] Mustapa A, Justine M, Mohd Mustafah N, Jamil N, Manaf H. Postural Control and Gait Performance in the Diabetic Peripheral Neuropathy: A Systematic Review. Biomed Res Int. 2016;2016:9305025. doi: 10.1155/2016/9305025. Epub 2016 Jul 20. PMID 27525281
- [Background] Oppenheim U, Kohen-Raz R, Alex D, Kohen-Raz A, Azarya M. Postural characteristics of diabetic neuropathy. Diabetes Care. 1999 Feb;22(2):328-32. doi: 10.2337/diacare.22.2.328. PMID 10333953
- [Background] Thukral N, Kaur J, Malik M. A Systematic Review and Meta-analysis on Efficacy of Exercise on Posture and Balance in Patients Suffering from Diabetic Neuropathy. Curr Diabetes Rev. 2021;17(3):332-344. doi: 10.2174/1573399816666200703190437. PMID 32619175
- [Background] Ledin T, Odkvist LM, Vrethem M, Moller C. Dynamic posturography in assessment of polyneuropathic disease. J Vestib Res. 1990-1991;1(2):123-8. PMID 1670145
- [Background] Dingwell JB, Ulbrecht JS, Boch J, Becker MB, O'Gorman JT, Cavanagh PR. Neuropathic gait shows only trends towards increased variability of sagittal plane kinematics during treadmill locomotion. Gait Posture. 1999 Sep;10(1):21-9. doi: 10.1016/s0966-6362(99)00016-8. PMID 10469938
- [Background] Grewal GS, Sayeed R, Schwenk M, Bharara M, Menzies R, Talal TK, Armstrong DG, Najafi B. Balance rehabilitation: promoting the role of virtual reality in patients with diabetic peripheral neuropathy. J Am Podiatr Med Assoc. 2013 Nov-Dec;103(6):498-507. doi: 10.7547/1030498. PMID 24297986
- [Background] Najafi B, Crews RT, Wrobel JS. A novel plantar stimulation technology for improving protective sensation and postural control in patients with diabetic peripheral neuropathy: a double-blinded, randomized study. Gerontology. 2013;59(5):473-80. doi: 10.1159/000352072. Epub 2013 Jul 16. PMID 23860103
- [Background] Morrison S, Colberg SR, Parson HK, Vinik AI. Relation between risk of falling and postural sway complexity in diabetes. Gait Posture. 2012 Apr;35(4):662-8. doi: 10.1016/j.gaitpost.2011.12.021. Epub 2012 Jan 23. PMID 22269128
- [Background] Kelly C, Fleischer A, Yalla S, Grewal GS, Albright R, Berns D, Crews R, Najafi B. Fear of falling is prevalent in older adults with diabetes mellitus but is unrelated to level of neuropathy. J Am Podiatr Med Assoc. 2013 Nov-Dec;103(6):480-8. doi: 10.7547/1030480. PMID 24297984
- [Background] Bouhassira D, Attal N, Alchaar H, Boureau F, Brochet B, Bruxelle J, Cunin G, Fermanian J, Ginies P, Grun-Overdyking A, Jafari-Schluep H, Lanteri-Minet M, Laurent B, Mick G, Serrie A, Valade D, Vicaut E. Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain. 2005 Mar;114(1-2):29-36. doi: 10.1016/j.pain.2004.12.010. Epub 2005 Jan 26. PMID 15733628
- [Background] Bennett M. The LANSS Pain Scale: the Leeds assessment of neuropathic symptoms and signs. Pain. 2001 May;92(1-2):147-57. doi: 10.1016/s0304-3959(00)00482-6. PMID 11323136
- [Background] Harden RN. Chronic neuropathic pain. Mechanisms, diagnosis, and treatment. Neurologist. 2005 Mar;11(2):111-22. doi: 10.1097/01.nrl.0000155180.60057.8e. PMID 15733333